CLINICAL TRIAL: NCT04872790
Title: A Dose-Finding Phase Ib Study of the Oral BCL-2 Inhibitor Venetoclax (ABT-199) in Combination With Standard Induction Therapy, Dasatinib and Prednisone (and Rituximab in CD20+ Patients), in Adult Patients With Newly Diagnosed and Relapsed Philadelphia Chromosome Positive (Ph+) ALL and Ph+ MPAL
Brief Title: Venetoclax, Dasatinib, Prednisone, Rituximab and Blinatumomab for the Treatment of Newly Diagnosed or Relapsed Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia or Mixed Phenotype Acute Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: AbbVie (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jessica Leonard, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022691; NCI-2021-01791 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022691 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-03-19; First posted 2021-05-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: B Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Mixed Phenotype Acute Leukemia; Recurrent B Acute Lymphoblastic Leukemia; Recurrent Mixed Phenotype Acute Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia, Biphenotypic, Acute | interventions — Dasatinib; Methotrexate; merphos; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; venetoclax; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Biopsy; Spinal Puncture; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (prednisone, dasatinib, venetoclax, rituximab) (Experimental): See detailed description
  Interventions: Drug: Dasatinib; Drug: Methotrexate; Drug: Prednisone; Biological: Rituximab; Drug: Venetoclax; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Lumbar Puncture; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel; BMS354825
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima; BI-695500; BI695500; Blitzima; IDEC 102; IDEC102; PF05280586; Ritemvia; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto; ABT 199; GDC0199
Biological: Blinatumomab — Given IV
  Other Names: 853426-35-4; AMG 103, Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI-538; MEDI538; MT103; AMG-103; AMG103; MEDI 538; MT 103; MT-103
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; spinal tap
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase Ib trial studies the effects of venetoclax in combination with dasatinib, prednisone, rituximab and blinatumomab in treating patients with Philadelphia chromosome positive acute lymphoblastic leukemia (ALL) that is newly diagnosed or that has come back (relapsed). Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Anti-inflammatory drugs, such as prednisone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Rituximab and blinatumomab are monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Giving venetoclax in combination with dasatinib, prednisone, and rituximab and blinatumomab may help treat patients with newly diagnosed or relapsed Philadelphia chromosome positive acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine amaximum tolerated dose (MTD) and a subsequently recommended phase II dose (RP2D) of venetoclax in combination with dasatinib.

II. Evaluate the safety of venetoclax in combination with dasatinib by assessing the frequency, type, and severity of adverse events.

SECONDARY OBJECTIVES:

I. Assess preliminary response to treatment based on minimal residual disease (MRD) negativity after venetoclax plus dasatinib induction and venetoclax, dasatinib, and blinatumomab consolidation.

II. Estimate progression-free and overall survival.

EXPLORATORY OBJECTIVES:

I. Evaluate the distribution of BCR-ABL fusion sub-types. II. Assess changes in BCL-family dependence. III. Presence of co-occurring leukemia-specific mutations. IV. Assess ex vivo sensitivity to venetoclax and dasatinib using inhibitor plates and colorimetric cell viability (MTS) assay.

V. Evaluate differences between two methods of detecting MRD for B ALL/mixed phenotype acute leukemia (MPAL): Real-time quantitative polymerase chain reaction (RQ PCR) analysis of BCR-ABL and next generation (NextGen) sequencing.

VI. Assess response after consolidation with blinatumomab, venetoclax, and dasatinib.

OUTLINE: This is dose-escalation study of venetoclax.

INDUCTION PHASE CYCLE 1: Patients receive prednisone orally (PO) once daily (QD) on days -6 to 21 and rapid taper from days 22-28, dasatinib PO QD days 1-28, venetoclax PO QD days 3-28 or days 3-21, rituximab (for CD20+ patients) intravenously (IV) on days 8 and 15, and methotrexate intrathecally (IT) once during week 1 and once during week 3 as prophylaxis or once a week (QW) as therapy in the absence of disease progression or unacceptable toxicity.

INDUCTION PHASE CYCLES 2-3: Patients receive dasatinib PO QD days 1-28, venetoclax PO QD on days 1-28 or 1-21, rituximab (for CD20+ patients) IV on days 1 and 15, and methotrexate IT on days 1 and 15. Treatment repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with clinical benefit may continue to receive treatment for up to 12 months per the discretion of the physician.

CONSOLIDATION CYCLES 4-7 (ALL PATIENTS ONLY): Patients receive blinatumomab IV on days 1-28. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients continue to receive dasatinib PO QD and venetoclax PO QD as taken in cycles 1-3 and, if clinically indicated, methotrexate IT on day 1. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy and aspiration, lumbar puncture, and blood sample collection throughout the study

MAINTENANCE THERAPY CYCLES 8+: Patients receive dasatinib PO QD and venetoclax PO QD as in consolidation cycles and, if clinically indicated, methotrexate IT on day 1 of cycles 8 and 9. Cycles repeat every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 12 weeks for up to 1 year.

Additionally, patients undergo bone marrow biopsy and aspiration, lumbar puncture, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 4 weeks and then for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have diagnosis of B acute lymphoblastic leukemia harboring the t(9;22) translocation (Philadelphia chromosome positive acute lymphoblastic leukemia [Ph+ ALL]) or Ph+ mixed phenotype acute leukemia (MPAL)) confirmed according to criteria.
* Diagnosis of MPAL will only be considered for enrollment during the dose finding period. Participants with MPAL will be enrolled for induction therapy only
* All individuals must have a bone marrow biopsy completed during the screening period. Patients with central nervous system (CNS) disease will be included
* Expression of CD19 by flow cytometry on bone marrow, if individual has received prior chimeric antigen receptor (CAR) T therapy. If CD19 negative, enrollment may be considered for induction treatment only
* Newly diagnosed subjects must have received no prior treatment for their ALL with the exception of steroids (prednisone, dexamethasone), hydrea or IT methotrexate. Individuals may receive pre-treatment with steroids during the screening phase prior to enrollment
* Individuals with relapsed disease may not have had prior treatment with dasatinib, however treatment with other tyrosine kinases is permitted
* At least 3 half-lives must have passed before cycle 1 day 1 (C1D1) for participants that have used strong CYP3A inhibitors (such as fluconazole, ketoconazole and clarithromycin) prior to enrollment
* At least 3 half-lives must have passed before cycle 1 day 3 (C1D3) for participants that have used moderate CYP3A inhibitors (such as fluconazole, ketoconazole and clarithromycin), strong or moderate CYP3A inducers (such as rifampin, carbamazepine, phenytoin, and St. John's wort), P-glycoprotein (P-gp) inhibitors, or warfarin prior to enrollment
* At least 4 weeks must have passed before (C1D3) for participants that have recently received a live vaccine
* Age >= 18 years. All participants irrespective of their gender identity and members of all races and ethnic groups will be included
* Eastern Cooperative Oncology Group (ECOG) status =< 2
* Must be able to take oral medication
* Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN)

  * Unless considered due to leukemic organ involvement
* Alanine aminotransferase (ALT) < 2.5 x ULN

  * Unless considered due to leukemic involvement
* Total bilirubin < 1.5 x ULN

  * Unless considered due to leukemic organ involvement
  * Note: subjects with Gilbert's Syndrome may have a bilirubin > 1.5 x ULN per discussion between the investigator and AbbVie medical monitor
* Subject must have adequate renal function as demonstrated by a calculated creatinine clearance >= 50 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft-Gault formula
* Persons of childbearing potential must have a negative serum or urine pregnancy test (sensitivity < 25 IU human chorionic gonadotropin [HCG]/L) within 72 hours prior to the start of the study drug
* Persons of reproductive potential must agree to use a highly effective method of contraception throughout treatment and for at least 4 weeks after study drug is stopped. Persons of childbearing potential and persons with a sexual partner of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy
* Normal corrected QT Formula (QTcF) interval on screening electrocardiogram (EKG) (< 450 ms regardless of sex)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* For newly diagnosed subjects: who have received treatment with cytotoxic chemotherapy, radiotherapy or immunotherapy for their ALL/MPAL, or prior dasatinib treatment. For relapsed subjects: prior dasatinib treatment (however treatment with other tyrosine kinase inhibitors [TKIs] is permitted)
* Subjects who have received any investigational agents or subjects who are taking investigational or commercial agents or therapies with the intent to treat the subject's malignancy within seven days or three half-lives of enrollment (i.e. initiation of dasatinib)
* Subjects with chronic myelogenous leukemia (CML) in myeloid blast crisis, Ph+ acute myeloid leukemia (AML) or acute leukemia lineage that cannot be classified based on existing criteria (e.g., from the World Health Organization [WHO] or International Consensus Classification [ICC])
* Subjects with clinically serious infections as determined by the provider requiring ongoing antibiotic therapy. This does not include antibiotic treatment for neutropenic fever
* Individuals with a pleural or pericardial effusion of any grade
* Subjects with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib or other agents used in the study
* Subjects who have undergone stem cell transplant must be at least 100 days after transplant, and without active treatment for graft versus host disease (GVHD) other than topical medications
* Subjects with uncontrolled cardiac illness including but not limited to, symptomatic congestive heart failure, unstable angina pectoris, clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes), or pulmonary hypertension
* Subjects with diagnosed congenital prolonged QT syndrome
* Pregnant persons are excluded from this study because dasatinib is a pregnancy category D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with dasatinib, breastfeeding should be discontinued if the mother is treated with dasatinib. These potential risks may also apply to venetoclax for which the pregnancy category and risks to the fetus are unknown
* Participant is seropositive with human immunodeficiency virus (HIV) or has active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).

  * HIV-infected individuals on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
  * For individuals with evidence of chronic HBV infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Individuals with a history of HCV infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Subjects with invasive malignancy over the previous year except treated early stage carcinomas of the skin, completely resected intraepithelial carcinoma of the cervix, completely resected papillary thyroid and follicular thyroid cancers, and localized prostate cancer treated with curative intent with surgery or radiation
* Subjects with any gastrointestinal condition which would lead to inability to absorb an oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2026-12-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | At day 32 (after 30 days of combination therapy)
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications. In order to be declared a dose-limiting toxicity, an adverse experience must be determined related (definitely, probably, or possibly) to study drug. Point estimates and 95% exact confidence intervals will be reported for all patients in the safety set as well as in subgroups defined by whether or not a patient received blinatumomab consolidation therapy.
Incidence of adverse events | Up to 90 days after last dose of study drug
  Adverse events will be graded and categorized according to the Common Terminology Criteria for Adverse Events version 5.0. Point estimates and 95% exact confidence intervals will be reported.

SECONDARY OUTCOMES:
Rate of complete molecular remission (CMR) | Up to completion of cycle 3 (1 cycle = 28 days)
Duration of complete molecular response (CMR) | From date of CMR to date of molecular relapse, death or date of last follow-up, assessed up to 12 months after discontinuing study therapy
  The proportion of subjects with CMR as previously defined and its 95% exact confidence interval will be estimated using the efficacy analysis set. Will be estimated using the Kaplan-Meier method along with 95% exact confidence interval.
Progression-free survival | From first dose of dasatinib to relapse, disease progression, death, date of last follow-up, assessed up to 12 months after discontinuing study therapy
  Will be estimated using the Kaplan-Meier method along with 95% exact confidence interval.
Overall survival | From first dose of dasatinib to death from any cause, assessed up to 12 months after discontinuing study therapy
  Will be estimated using the Kaplan-Meier method along with 95% exact confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica T Leonard, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States